CLINICAL TRIAL: NCT03449862
Title: Effect of Clinical Decision Rules, Patient Cost and Malpractice Information on Clinician Brain CT Image Ordering: a Randomized Controlled Trial
Brief Title: Key Information Can Influence Clinician Ordering of Brain CTs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clemson University (Other)
Collaborators: Prisma Health-Upstate (Other); Emory University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Pro00054122
Record Dates: First submitted 2018-02-14; First posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Clinical Decision-Making

STUDY DESIGN:
Intervention Model Description: Multi-center, double-blinded simulation-based randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Electronic web-based simulation study with built-in randomization tool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LEGAL-COST (Experimental): Clinicians were first presented malpractice case law summary information (which suggests clinician not likely to be sued for not ordering CT scan) then patient out-of-pocket cost information for brain CT image (which provides them insight into what the patient is likely to pay for the test)
  Interventions: Other: Simulation-based clinical decision on brain CT ordering
- COST-LEGAL (Active Comparator): Clinicians were first presented with patient out-of-pocket cost information for brain CT image (which provides them insight into what the patient is likely to pay for the test) then malpractice case law summary information (which suggests clinician not likely to be sued for not ordering CT scan)
  Interventions: Other: Simulation-based clinical decision on brain CT ordering

INTERVENTIONS:
Other: Simulation-based clinical decision on brain CT ordering — Clinicians asked to make decision on medical imaging for their simulated patient after presentation of clinical case then additional information. At each presentation of new information the clinician may modify their image order.

SUMMARY:
The frequency of head computed tomography (CT) imaging for mild head trauma patients has raised safety and cost concerns. Validated clinical decision rules exist in the published literature and on-line sources to guide medical image ordering but are often not used by emergency department (ED) clinicians. Using simulation, we explored whether the presentation of a clinical decision rule (i.e. Canadian CT Head Rule - CCHR), findings from malpractice cases related to clinicians not ordering CT imaging in mild head trauma cases, and estimated patient out-of-pocket cost might influence clinician brain CT ordering. Understanding what type and how information may influence clinical decision making in the ordering advanced medical imaging is important in shaping the optimal design and implementation of related clinical decision support systems.

DETAILED DESCRIPTION:
Multi-center, double-blinded simulation-based randomized controlled trial. Following standardized clinical vignette presentation, clinicians made an initial imaging decision for the patient. This was followed by additional information on decision support rules, malpractice outcome review, and patient cost; each with opportunity to modify their initial order. The malpractice and cost information differed by assigned group to test the any temporal relationship. The simulation closed with a second vignette and an imaging decision.

ELIGIBILITY:
Inclusion Criteria:

* Clinician (physician, nurse practitioner, physician assistant) licensed to deliver health care.
* Actively employed to deliver health care in the emergency department of Greenville health System (South Carolina) or Emory University (Georgia)

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2018-02-13 (Actual)

PRIMARY OUTCOMES:
brain CT medical image order | 30 days
  At each decision point clinician asked to decide on which image to order for patient among three choices:
  * CT Head without/with contrast
  * CT Head without contrast
  * No medical imaging

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W. Gimbel, PHD, Principal Investigator — Clemson University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gimbel RW, Pirrallo RG, Lowe SC, Wright DW, Zhang L, Woo MJ, Fontelo P, Liu F, Connor Z. Effect of clinical decision rules, patient cost and malpractice information on clinician brain CT image ordering: a randomized controlled trial. BMC Med Inform Decis Mak. 2018 Mar 12;18(1):20. doi: 10.1186/s12911-018-0602-1. PMID 29530029

DOCUMENTS (3):
  • Study Protocol (2016-11-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT03449862/Prot_000.pdf
  • Informed Consent Form (2016-05-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT03449862/ICF_001.pdf
  • Statistical Analysis Plan (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT03449862/SAP_002.pdf